CLINICAL TRIAL: NCT07300124
Title: Outcome of Direct Pulp Capping and Partial Pulpotomy in Reversible Pulpitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pankaj Sangwan
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Reversible Pulpitis; Extremely Deep Caries
Keywords: Partial Pulpotomy; Direct pulp capping
MeSH Terms: interventions — Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Pulp Capping in Reversible Pulpitis (Experimental): Direct Pulp Capping will be performed on carious pulp exposure after establishing a clinical diagnosis of symptomatic reversible pulpitis based on history of pain exacerbated by cold stimuli and subsides on removal of stimuli compared to normal teeth and which is reproducible using cold testing.
  Interventions: Procedure: Direct pulp capping with MTA
- Partial Pulpotomy in Reversible Pulpitis (Active Comparator): Partial Pulpotomy will be performed on carious pulp exposure after establishing a clinical diagnosis of symptomatic reversible pulpitis based on history of pain exacerbated by cold stimuli and subsides on removal of stimuli compared to normal teeth and which is reproducible using cold testing.
  Interventions: Procedure: Partial Pulpotomy in Reversible Pulpitis

INTERVENTIONS:
Procedure: Partial Pulpotomy in Reversible Pulpitis — Procedure/Surgery: Outcome of Partial Pulpotomy in teeth with clinical signs indicative of Reversible Pulpitis with extremely deep caries.
  After caries removal and pulp exposure , 2-3 mm of pulp tissue will be amputated and the pulpal wound irrigated with 3% NaOCl. Bleeding will be controlled by placing a cotton pellet soaked in 3% NaOCl over the pulpal wound for 2-3 minutes, repeated if required. This will be followed by capping with a 2-3 mm layer of MTA in both the groups. A layer of RMGIC will then be placed over the MTA, and the tooth will be permanently restored with composite resin.
  Arms: Partial Pulpotomy in Reversible Pulpitis
Procedure: Direct pulp capping with MTA — Outcome of direct pulp capping in teeth with clinical signs indicative of reversible pulpitis.
  After caries removal and pulp exposure pulpal wound will be irrigated with 3% NaOCl, and bleeding will be controlled by placing a cotton pellet soaked with 3% NaOCl over the pulpal wound for 2 to 3 minutes and will be repeated if required. Followed by capping with MTA, a layer of RMGIC will be placed over the MTA. Then the tooth will be permanently restored with composite resin.
  Arms: Direct Pulp Capping in Reversible Pulpitis

SUMMARY:
AIM: -The aim of the study is to compare the outcome of Direct Pulp Capping and Partial Pulpotomy in mature permanent teeth with Reversible Pulpitis OBJECTIVES: - Primary Objective: to compare the difference in clinical and radiographic outcome of direct pulp capping and partial pulpotomy in mature permanent teeth with Reversible Pulpitis. Secondary objective: To evaluate and compare postoperative pain after Direct Pulp Capping and Partial Pulpotomy in teeth with Reversible Pulpitis STUDY GROUPS: - Subjects of age group 15 to 40 years will be included and divided into two groups

1. Direct Pulp Capping in Permanent mature molars with Reversible Pulpitis
2. Partial Pulpotomy in Permanent mature molars with Reversible Pulpitis

DETAILED DESCRIPTION:
TITLE: Outcome of Direct Pulp Capping and Partial Pulpotomy in Reversible Pulpitis It aims to answer does outcome of direct pulp capping and partial pulpotomy differ in mature permanent teeth with extremely deep caries with reversible pulpitis. P (Population) - Mature permanent mandibular molars with extremely deep caries and clinical signs of reversible pulpitis. I (Intervention) -Direct Pulp Capping in teeth with Reversible Pulpitis. C (Comparison) -Partial Pulpotomy in teeth with Reversible Pulpitis. O (Outcome) -Assessment of clinical & radiographic success at 6 and 12 months follow up -Assessment of pain experience at baseline, post-operatively every 24 hours for 1 week In extremely deep lesions, the dental pulp is often inflamed or at risk of microbial contamination, therefore requiring timely and precise intervention in order to preserve pulp vitality. In such cases, the removal of the superficial 2-3 mm of inflamed pulp tissue can help maintain the health of the remaining pulpal tissue. Duncan and other researchers have emphasized the importance of assessing both caries depth and pulpal status for deciding the effective treatment plan. Although numerous studies have investigated the outcomes of Direct Pulp Capping (DPC) and Partial Pulpotomy separately & have included cases based on caries depth & pulpal status, such as reversible pulpitis. However, there remains a notable lack of comparative clinical studies directly evaluating partial pulpotomy and direct pulp capping under standardized conditions involving extremely deep carious lesions with pulpal status as reversible pulpitis. Hence, this clinical trial aims to assess and compare the clinical and radiographic outcome of Direct Pulp Capping and Partial Pulpotomy in extremely deep caries with reversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 15-40 years.
2. Mature permanent mandibular molars with extremely deep caries on radiograph, giving positive response to pulp sensibility test.
3. Pulpal bleeding can be controlled within 10 minutes
4. Patients having normal periapical status with periapical index (PAI) score ≤ 2
5. Periodontally healthy teeth
6. Positive response to pulp sensibility test

Exclusion Criteria:

1. Non restorable teeth
2. Negative response to vitality testing
3. Presence of sinus tract or soft tissue swelling
4. Absence of deep carious lesions radiographically
5. Radiographic signs of internal or external root resorption
6. Patient had moderate to severe pain, but preferred root canal treatment
7. Presence of sound dentin over pulp and pulp not exposed intraoperatively
8. Pulp haemorrhage could not be arrested within 10 minutes.
9. Necrotic pulp evident upon exposure
10. Pregnant women
11. Absence of antagonist teeth
12. Intake of antibiotics in last 30 days

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Success rate at 1 year | Baseline to 12 months
  Criteria for success:-
  Clinical:
  1. Absence of signs and symptoms of spontaneous pain or pain on stimulus and discomfort except for the first few days after treatment.
  2. No tenderness to palpation or percussion and the tooth is functional.
  3. Normal mobility and probing pocket depth.
  4. Absence of associated soft tissue swelling, sinus or fistula. Radiographic: -
  1. Absence of any periapical or interradicular radiolucency. 2. Complete radiographic healing (PAI score 1 or 2 acc. to Ostravik et al). 3. Absence of internal and external root resorption Tooth will be considered successful when all the above parameters are met.

SECONDARY OUTCOMES:
Postoperative Pain | Baseline and at 24 hours, Day 2, Day 3, Day 4, Day 5, Day 6 and Day 7 after the treatment
  Post Operative Pain- To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score100 means maximum pain. To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score 100 means maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Pankaj Sangwan, MDS, Principal Investigator — PGIDS, Rohtak, Haryana 124001
Locations (1):
- PGIDS Rohtak, Rohtak, Haryana, India